CLINICAL TRIAL: NCT00753272
Title: Observer-blind Superior Efficacy Trial With GlaxoSmithKline Biologicals' Influenza Vaccine GSK2186877A in Elderly Subjects
Brief Title: Trial to Evaluate the Efficacy of GSK Biologicals' Influenza Vaccine GSK2186877A in Adults 65 Year of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 106372
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2017-08

CONDITIONS: Influenza
Keywords: Efficacy; Influenza Vaccines; Influenza; Vaccine; Elderly
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- FluNG Group (Experimental): subjects received 2 doses (1 dose per season) of FluNG vaccine during the Northern Hemisphere (NH) vaccination periods. One dose at Day 0 of the Year 1 and one dose at Day 0 of the Year 2 (= Day 365 Year 1).
  Interventions: Biological: GSK Bio's influenza vaccine GSK2186877A
- Fluarix Group (Active Comparator): subjects received 2 doses (1 dose per season) of Fluarix™ vaccine during the Northern Hemisphere (NH) vaccination periods. One dose at Day 0 of the Year 1 and one dose at Day 0 of the Year 2 (= Day 365 Year 1).
  Interventions: Biological: Fluarix TM

INTERVENTIONS:
Biological: GSK Bio's influenza vaccine GSK2186877A — IM administration, two times one annual dose, 3 different lots will be tested
  Arms: FluNG Group
Biological: Fluarix TM — IM administration, two times one annual dose
  Arms: Fluarix Group

SUMMARY:
The purpose of this study is to evaluate the efficacy of GlaxoSmithKline Biologicals' influenza vaccine GSK2186877A in adults 65 year of age and older. The study design is divided in two surveillance phases: one passive phase along the study during the influenza season and one active surveillance phase during the influenza peak season.

DETAILED DESCRIPTION:
This Protocol Posting has been updated according to Protocol Amendment 3, Sep 2009.

After the analyses for this study were completed, questions arose regarding the integrity of study data from a single study site in Romania, which enrolled 102 subjects in the trial. Because evaluation of data from this site did not reveal irregularities when compared with overall study data and because GSK has no current plans to use the data from the study in support of any regulatory filings, they were not excluded from the analyses reflected in this results summary.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A man or woman aged 65 years or older at the time of the vaccination.
* Written informed consent obtained from the subject.
* Subjects with residence status allowing free mixing with general community.

Exclusion Criteria:

* Bedridden subjects
* Previous vaccination against influenza since February 2008.
* Previous vaccination in the last three years with an investigational adjuvanted candidate seasonal or pandemic influenza vaccine.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Any contra-indication to intramuscular administration of the influenza vaccines.
* History of hypersensitivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine including egg and chicken protein.
* Acute disease at the time of enrolment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e. Oral temperature <37.5°C (99.5°F).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 43695 (Actual)
Dates: Start 2008-09-15 (Actual); Primary Completion 2010-06-18 (Actual); Study Completion 2011-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (217):
- United States (54):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Crystal River, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Inverness, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Camillus, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Salisbury, North Carolina
  - GSK Investigational Site, Tabor City, North Carolina
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Grove City, Pennsylvania
  - GSK Investigational Site, Jefferson Hills, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Upper Saint Clair, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, North Myrtle Beach, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Marshfield, Wisconsin
- Belgium (16):
  - GSK Investigational Site, Anthée
  - GSK Investigational Site, Deinze
  - GSK Investigational Site, Dour
  - GSK Investigational Site, Drongen
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Gozée
  - GSK Investigational Site, Kerksken
  - GSK Investigational Site, Libramont
  - GSK Investigational Site, Linkebeek
  - GSK Investigational Site, Maldegem
  - GSK Investigational Site, Melsbroek
  - GSK Investigational Site, Merelbeke
  - GSK Investigational Site, Mettet
  - GSK Investigational Site, Natoye
  - GSK Investigational Site, Oostakker
  - GSK Investigational Site, Waarschoot
- Canada (12):
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, St-Romulad, Quebec
- Czechia (3):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Jaroměř
  - GSK Investigational Site, Pardubice
- Estonia (3):
  - GSK Investigational Site, Saku
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (28):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Anzin
  - GSK Investigational Site, Arras
  - GSK Investigational Site, Bécon-les-Granits
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Chambéry
  - GSK Investigational Site, Château-Gontier
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Écouflant
  - GSK Investigational Site, Grésy-sur-Aix
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Le Fousseret
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Montreuil-Juigné
  - GSK Investigational Site, Muret
  - GSK Investigational Site, Nieul-sur-Mer
  - GSK Investigational Site, Oignies
  - GSK Investigational Site, Orthez
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Segré
  - GSK Investigational Site, Seysses
  - GSK Investigational Site, Tiercé
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Vourey
- Germany (54):
  - GSK Investigational Site, Güglingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Messkirch, Baden-Wurttemberg
  - GSK Investigational Site, Rudersberg, Baden-Wurttemberg
  - GSK Investigational Site, Schwetzingen, Baden-Wurttemberg
  - GSK Investigational Site, Sinsheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Ketzin, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Bad Kreuznach, Hesse
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Brinkum/Stuhr, Lower Saxony
  - GSK Investigational Site, Duelmen, Lower Saxony
  - GSK Investigational Site, Koenigslutter, Lower Saxony
  - GSK Investigational Site, Rotenburg (Wümme), Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Ingelheim, Rhineland-Palatinate
  - GSK Investigational Site, Kallstadt, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Borna, Saxony
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freiberg, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Geringswalde, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Weißenberg, Saxony
  - GSK Investigational Site, Köthen, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Bad Bramstedt, Schleswig-Holstein
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Erfurt, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Mexico (4):
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Ecatepec de Morelos, State of Mexico
  - GSK Investigational Site, México
- Netherlands (3):
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Soest
  - GSK Investigational Site, Utrecht
- Norway (8):
  - GSK Investigational Site, Ålesund
  - GSK Investigational Site, Bekkestua
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Skien
  - GSK Investigational Site, Stavanger
- Poland (17):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Grodzisk Mazowiecki
  - GSK Investigational Site, Inowrocław
  - GSK Investigational Site, Iława
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lubartów
  - GSK Investigational Site, Oleśnica
  - GSK Investigational Site, Porąbka
  - GSK Investigational Site, Płock
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Tychy
  - GSK Investigational Site, Wroclaw
- Romania (7):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Brăila
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Galati
  - GSK Investigational Site, Pantelimon
  - GSK Investigational Site, Ploieşti
- Russia (3):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Yekaterinburg
- GSK Investigational Site, Taipei, Taiwan
- United Kingdom (4):
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Waterloo, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Ruiz-Palacios GM, Leroux-Roels G, Beran J, Devaster JM, Esen M, Launay O, McElhaney JE, van Essen GA, Benoit A, Claeys C, Dewe W, Durand C, Duval X, Falsey AR, Feldman G, Galtier F, Gervais P, Hwang SJ, McNeil S, Richardus JH, Trofa A, Oostvogels L; Influence65 study group. Immunogenicity of AS03-adjuvanted and non-adjuvanted trivalent inactivated influenza vaccines in elderly adults: A Phase 3, randomized trial and post-hoc correlate of protection analysis. Hum Vaccin Immunother. 2016 Dec;12(12):3043-3055. doi: 10.1080/21645515.2016.1219809. PMID 27690762
- [Derived] van Essen GA, Beran J, Devaster JM, Durand C, Duval X, Esen M, Falsey AR, Feldman G, Gervais P, Innis BL, Kovac M, Launay O, Leroux-Roels G, McElhaney JE, McNeil S, Oujaa M, Richardus JH, Ruiz-Palacios G, Osborne RH, Oostvogels L. Influenza symptoms and their impact on elderly adults: randomised trial of AS03-adjuvanted or non-adjuvanted inactivated trivalent seasonal influenza vaccines. Influenza Other Respir Viruses. 2014 Jul;8(4):452-62. doi: 10.1111/irv.12245. Epub 2014 Apr 4. PMID 24702710
- [Derived] McElhaney JE, Beran J, Devaster JM, Esen M, Launay O, Leroux-Roels G, Ruiz-Palacios GM, van Essen GA, Caplanusi A, Claeys C, Durand C, Duval X, El Idrissi M, Falsey AR, Feldman G, Frey SE, Galtier F, Hwang SJ, Innis BL, Kovac M, Kremsner P, McNeil S, Nowakowski A, Richardus JH, Trofa A, Oostvogels L; Influence65 study group. AS03-adjuvanted versus non-adjuvanted inactivated trivalent influenza vaccine against seasonal influenza in elderly people: a phase 3 randomised trial. Lancet Infect Dis. 2013 Jun;13(6):485-96. doi: 10.1016/S1473-3099(13)70046-X. Epub 2013 Mar 19. PMID 23518156
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 106372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106372 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were vaccinated during the pre-influenza season at Day 0, were contacted by phone during the surveillance period from mid November to the end of the influenza season (April-May) and were contacted by phone at Days 270 and 365 for the Year 1 influenza season 2008/2009 and the Year 2 influenza season 2009/2010.
Pre-assignment Details: For lot-to-lot consistency analyses after Dose 1 at Day 0 of the Year 1, FluNG Group was divided in 3 sub-groups: FluNG Lot 1 Group, FluNG Lot 2 Group and FluNG Lot 3 Group: subjects received 1 dose of FluNG vaccine Lot 1, 2 or 3 at Day 0 of the Year 1. They all received Dose 2 at Day 0 of the Year 2, again from 3 different lots.
Groups:
- Fluarix Group: subjects received 2 doses (1 dose per season) of Fluarix vaccine during the Northern Hemisphere (NH) vaccination periods. One dose at Day 0 of the Year 1 and one dose at Day 0 of the Year 2 (= Day 365 Year 1).
Period: Overall Study
Arm/Group | FluNG Group | Fluarix Group
Started | 21893 | 21802
Completed | 16911 | 16895
Not Completed | 4982 | 4907
Not completed — Adverse Event | 878 | 869
Not completed — Protocol Violation | 28 | 46
Not completed — Withdrawal by Subject | 2481 | 2407
Not completed — Lost to Follow-up | 491 | 497
Not completed — Other | 1104 | 1088

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluNG Group | Fluarix Group | Total
Number analyzed (Participants) | 21893 | 21802 | 43695
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.5 (6.09) | 73.5 (6.16) | 73.5 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12549 | 12422 | 24971
  Male | 9344 | 9380 | 18724

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Polymerase Chain Reaction (PCR)-Confirmed Influenza A and/or B Infection.
Description: Occurrence of PCR-confirmed influenza A and/or B infection, due to any matching or drift influenza strain relative to the vaccine strains (i.e. not emerging novel human influenza strain like H1N1v). PCR-confirmed influenza (PCI) was defined as an episode of influenza-like illness (ILI) occurring after the administration of the study vaccine for which a nasal and throat swab specimen yields influenza virus A and/or B by reverse transcription polymerase chain reaction (RT-PCR) analysis.
Time Frame: After the first dose during the corresponding surveillance period (from mid November 2008 to the end of April 2009 (end of influenza season))
Population: The One-Dose According-To-Protocol cohort for efficacy included eligible subjects from the One-Dose Total Vaccinated cohort (e.g. who complied with the protocol, with no elimination criteria assigned during the study), who had started their first surveillance period, who had not received a seasonal influenza vaccine not foreseen in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 21573 | 21482
Participants | 274 | 310

2. Primary Outcome: Serum Hemagglutination-inhibition (HI) Antibody Titers, Against Each of the 3 Vaccine Influenza Strains, in the FluNG Groups.
Description: Vaccine strains assessed were A/Brisbane/59/2077, A/Uruguay/716/2007 and B/Brisbane/3/2007. Titers were expressed as geometric mean titers calculated on all subjects in the lot-to-lot subset of subjects.
Time Frame: At Days 0 (pre-vaccination Dose 1) and 21 (post-vaccination Dose 1) of the first year (2008/2009) of the study
Population: The One-Dose According-To-Protocol immunogenicity cohort for the lot-to-lot consistency subset, which included all subjects from the One-Dose ATP cohort for immunogenicity included in the lot-to-lot subset.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- FluNG Lot 1 Group: subjects received 1 dose of FluNG vaccine Lot 1 at Day 0 of the Year 1. They received Dose 2 at Day 0 of the Year 2, again from lot 1. The vaccine was administered intramuscularly in the non-dominant deltoid.
- FluNG Lot 2 Group: subjects received 1 dose of FluNG vaccine Lot 2 at Day 0 of the Year 1. They received Dose 2 at Day 0 of the Year 2, again from lot 2. The vaccine was administered intramuscularly in the non-dominant deltoid.
- FluNG Lot 3 Group: subjects received 1 dose of FluNG vaccine Lot 3 at Day 0 of the Year 1. They received Dose 2 at Day 0 of the Year 2, again from lot 3. The vaccine was administered intramuscularly in the non-dominant deltoid.
Arm/Group | FluNG Lot 1 Group | FluNG Lot 2 Group | FluNG Lot 3 Group
Number analyzed (Participants) | 540 | 538 | 534
Titers
  A/Brisbane [Day 0]: number analyzed (Participants) | 539 | 536 | 532
  A/Brisbane [Day 0] | 15.9 [14.6 to 17.3] | 15.8 [14.5 to 17.2] | 15.8 [14.5 to 17.2]
  A/Brisbane [Day 21] | 82.3 [75.0 to 90.2] | 83.6 [76.0 to 92.0] | 93.4 [84.6 to 103.1]
  A/Uruguay [Day 0]: number analyzed (Participants) | 539 | 536 | 532
  A/Uruguay [Day 0] | 18.2 [16.5 to 20.2] | 17.8 [16.0 to 19.9] | 17.3 [15.6 to 19.2]
  A/Uruguay [Day 21] | 272.5 [243.0 to 305.6] | 287.5 [256.2 to 322.7] | 269.9 [239.9 to 303.6]
  B/Brisbane[Day 0]: number analyzed (Participants) | 539 | 536 | 532
  B/Brisbane[Day 0] | 94.2 [84.8 to 104.7] | 89.9 [80.6 to 100.3] | 87.1 [78.3 to 96.7]
  B/Brisbane[Day 21] | 652.4 [602.0 to 707.1] | 596.9 [552.2 to 645.3] | 601.7 [555.0 to 652.4]

3. Secondary Outcome: Number of Subjects Reporting Polymerase Chain Reaction (PCR)-Confirmed Influenza A and/or B Infection.
Description: as for outcome 1
Time Frame: During the whole surveillance period (from mid November 2008 to end of April 2009 and from mid November 2009 to end of April 2010)
Population: The According-To-Protocol cohort for efficacy included all eligible subjects from the Total Vaccinated cohort (e.g. who complied with the protocol, with no elimination criteria assigned during the study), who had started their first surveillance period, who had not received a seasonal influenza vaccine not foreseen in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 20579 | 20458
Participants | 262 | 296

4. Secondary Outcome: Number of Subjects Reporting Culture-confirmed Influenza A and/or B Infection.
Description: Occurrence of culture-confirmed influenza A and/or B infection, due to any matching or drift influenza strain relative to the vaccine strains (i.e. not emerging novel human influenza strain like H1N1v). Culture-confirmed influenza (CCI) was defined as an episode of ILI occurring after the administration of the study vaccine for which a nasal and throat swab specimen yields influenza virus A and/or B by viral culture analysis.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 20579 | 20458
Participants | 144 | 145

5. Secondary Outcome: Number of Subjects Reporting Pneumonia or Clinical Influenza After the First Dose of Vaccine.
Description: Clinical influenza= An ILI episode (with an ILI onset from the 15th of November until the end of the surveillance period) with at least simultaneously fever (oral temperature of ≥37.8 degrees Celsius) and cough.
  The influenza peak season = period during the study with the highest incidence of any matching or drift influenza strain relative to the vaccine strains (i.e. not emerging novel human influenza strain like H1N1v).
Time Frame: During the influenza peak season within the first surveillance period (the influenza peak season being defined per country, falling somewhere between mid November 2008 to end of April 2009)
Population: The One-Dose According-To-Protocol cohort for efficacy for peak season included all subjects from the One-Dose ATP cohort for efficacy who did not drop out from the study before the start of their first influenza peak season.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 21394 | 21337
Participants | 202 | 225

6. Secondary Outcome: Number of Subjects Reporting All-cause Death After the First Dose of Vaccine.
Description: The influenza peak season = period during the study with the highest incidence of any matching or drift influenza strain relative to the vaccine strains (i.e. not emerging novel human influenza strain like H1N1v).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 21394 | 21337
Participants | 63 | 88

7. Secondary Outcome: Number of Subjects Reporting Hospitalization Due to Respiratory Diseases After the First Dose of Vaccine
Description: Respiratory disease: A diagnosis of respiratory disease included: acute respiratory infections, other diseases of upper respiratory tract, pneumonia and influenza, chronic obstructive pulmonary disease and allied conditions, pneumoconioses and other lung diseases due to external agents, other diseases of respiratory system. In case the event has a fatal outcome, the diagnosis can also be confirmed by autopsy.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 21394 | 21337
Participants | 84 | 89

8. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Adverse Events (AEs) of Specific Interest Including Autoimmune Disease (AID).
Description: Adverse events of specific interest for safety monitoring are a subset of AEs that included both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
  Grade 3 = event that prevented normal everyday activities Related = event assessed by the investigator as causally related to the study vaccination
Time Frame: Within 365 days after the first dose (from Dose 1 at Day 0 up to Day 365 for the Year 2008/2009)
Population: The One-Dose Total Vaccinated cohort included all subjects with one vaccine administration documented during the first year of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 21893 | 21802
Participants
  Any AEs | 70 | 60
  Grade 3 AEs | 13 | 8
  Related AEs | 11 | 7

9. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Adverse Events (AEs) of Specific Interest Including Autoimmune Disease (AID).
Description: as for outcome 8
Time Frame: Within 365 days after the second dose (from Dose 1 at Day 0 up to Day 365 for the Year 2009/2010)
Population: The Two-Dose Total Vaccinated cohort included all subjects with one vaccine administration documented in each year of the study
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 17070 | 17071
Participants
  Any AEs | 35 | 40
  Grade 3 AEs | 9 | 6
  Related AEs | 2 | 0

10. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Adverse Events (AEs) of Specific Interest Including Autoimmune Disease (AID).
Description: as for outcome 8
Time Frame: During the entire study period (during the 365 days of follow-up after each vaccination at Year 2008/2009 and Year 2009/2010)
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 21893 | 21802
Participants
  Any AEs | 103 | 99
  Grade 3 AEs | 22 | 14
  Related AEs | 13 | 7

11. Secondary Outcome: Number of Subjects Reporting Any and Related to Vaccination Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
  Related = event assessed by the investigator as causally related to the study vaccination
Time Frame: as for outcome 10
Population: The Total Vaccinated cohort included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 21893 | 21802
Participants
  Any SAEs | 4071 | 4066
  Related SAEs | 9 | 6

12. Secondary Outcome: Number of Subjects Reporting Any and Severe (Grade 3) Solicited Local Symptoms.
Description: Solicited local symptoms assessed were ecchymosis, pain, redness and swelling. Any = incidence of a particular symptom regardless of intensity grade. Grade 3 pain = considerable pain at rest that prevented normal everyday activities. Grade 3 ecchymosis/redness/swelling = ecchymosis/redness/swelling above 100 millimeter
Time Frame: During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Population: The One-Dose Total Vaccinated cohort for the safety subset included all subjects with at least one vaccine administration documented during the first year of the study and included in the safety subset.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 2988 | 2968
Participants
  Any ecchymosis | 40 | 18
  Ecchymosis > 100 mm | 0 | 0
  Any pain | 1225 | 477
  Grade 3 pain | 4 | 3
  Any redness | 240 | 66
  Redness > 100 mm | 6 | 3
  Any swelling | 189 | 40
  Swelling > 100 mm | 4 | 0

13. Secondary Outcome: Number of Days With Any Grade of Solicited Local Symptoms
Description: Solicited local symptoms assessed were ecchymosis, pain, redness and swelling
Time Frame: During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Population: as for outcome 12
Measure: Mean (Full Range); unit: Days
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 1221 | 476
Days
  Ecchymosis: number analyzed (Participants) | 39 | 18
  Ecchymosis | 3.6 [1.0 to 7.0] | 4.0 [1.0 to 7.0]
  Pain | 2.5 [1.0 to 7.0] | 2.1 [1.0 to 7.0]
  Redness: number analyzed (Participants) | 237 | 63
  Redness | 2.9 [1.0 to 7.0] | 2.5 [1.0 to 7.0]
  Swelling: number analyzed (Participants) | 186 | 40
  Swelling | 2.9 [1.0 to 7.0] | 2.0 [1.0 to 7.0]

14. Secondary Outcome: Number of Subjects Reporting Any and Severe (Grade 3) Solicited Local Symptoms
Description: as for outcome 12
Time Frame: During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Population: The Two-Dose Total Vaccinated cohort for the safety subset included all subjects with at least one vaccine administration documented in each year of the study and included in the safety subset.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 2441 | 2488
Participants
  Any ecchymosis | 39 | 31
  Ecchymosis > 100 mm | 1 | 0
  Any pain | 998 | 440
  Grade 3 pain | 13 | 7
  Any redness | 212 | 54
  Redness > 100 mm | 4 | 2
  Any swelling | 173 | 38
  Swelling > 100 mm | 3 | 0

15. Secondary Outcome: Number of Days With Any Grade of Solicited Local Symptoms.
Description: Solicited local symptoms assessed were ecchymosis, pain, redness and swelling.
Time Frame: During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Population: as for outcome 14
Measure: Mean (Full Range); unit: Days
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 995 | 431
Days
  Ecchymosis: number analyzed (Participants) | 28 | 22
  Ecchymosis | 2.8 [1.0 to 7.0] | 3.6 [1.0 to 7.0]
  Pain | 2.5 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Redness: number analyzed (Participants) | 202 | 46
  Redness | 2.8 [1.0 to 7.0] | 2.6 [1.0 to 7.0]
  Swelling: number analyzed (Participants) | 162 | 25
  Swelling | 2.5 [1.0 to 7.0] | 2.7 [1.0 to 7.0]

16. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Solicited General Symptoms
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, shivering and temperature (defined as oral temperature equal to or above (≥) 38.0 degrees Celsius). Any = incidence of a particular symptom regardless of intensity grade or relationship to vaccination. Grade 3 = general symptom which prevented normal everyday activities. Related = general symptom assessed by the investigator as causally related to the study vaccination. Grade 3 temperature = oral temperature ≥39.0°C - ≤ 40.0°C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 2986 | 2968
Participants
  Any arthralgia | 391 | 239
  Grade 3 arthralgia | 11 | 5
  Related arthralgia | 285 | 163
  Any fatigue | 646 | 417
  Grade 3 fatigue | 20 | 15
  Related fatigue | 494 | 295
  Any gastrointestinal | 197 | 165
  Grade 3 gastrointestinal | 6 | 4
  Related gastrointestinal | 132 | 82
  Any headache | 474 | 333
  Grade 3 headache | 8 | 4
  Related headache | 341 | 213
  Any myalgia | 547 | 302
  Grade 3 myalgia | 14 | 11
  Related myalgia | 412 | 203
  Any shivering | 245 | 80
  Grade 3 shivering | 12 | 2
  Related shivering | 185 | 49
  Temperature >= 38.0°C | 72 | 20
  Temperature >= 39.0°C - <=40.0°C | 5 | 2
  Related temperature | 51 | 14

17. Secondary Outcome: Number of Days With Any Grade of Solicited General Symptoms
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, shivering and temperature.
Time Frame: During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Population: as for outcome 12
Measure: Mean (Full Range); unit: Days
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 642 | 417
Days
  Arthralgia: number analyzed (Participants) | 388 | 239
  Arthralgia | 2.8 [1.0 to 7.0] | 2.9 [1.0 to 7.0]
  Fatigue | 2.5 [1.0 to 7.0] | 2.7 [1.0 to 7.0]
  Gastrointestinal: number analyzed (Participants) | 195 | 164
  Gastrointestinal | 2.2 [1.0 to 7.0] | 2.2 [1.0 to 7.0]
  Headache: number analyzed (Participants) | 472 | 332
  Headache | 2.2 [1.0 to 7.0] | 2.3 [1.0 to 7.0]
  Myalgia: number analyzed (Participants) | 544 | 301
  Myalgia | 2.3 [1.0 to 7.0] | 2.3 [1.0 to 7.0]
  Shivering: number analyzed (Participants) | 244 | 80
  Shivering | 1.6 [1.0 to 7.0] | 2.1 [1.0 to 7.0]
  Temperature: number analyzed (Participants) | 59 | 16
  Temperature | 1.4 [1.0 to 7.0] | 1.3 [1.0 to 4.0]

18. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related Solicited General Symptoms.
Description: as for outcome 16
Time Frame: During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 2436 | 2489
Participants
  Any arthralgia | 258 | 176
  Grade 3 arthralgia | 10 | 4
  Related arthralgia | 169 | 90
  Any fatigue | 457 | 318
  Grade 3 fatigue | 8 | 6
  Related fatigue | 307 | 169
  Any gastrointestinal | 137 | 124
  Grade 3 gastrointestinal | 5 | 8
  Related gastrointestinal | 71 | 46
  Any headache | 342 | 237
  Grade 3 headache | 10 | 4
  Related headache | 219 | 119
  Any myalgia | 380 | 209
  Grade 3 myalgia | 11 | 6
  Related myalgia | 261 | 117
  Any shivering | 189 | 88
  Grade 3 shivering | 11 | 6
  Related shivering | 127 | 44
  Temperature >= 38.0°C | 52 | 25
  Temperature >= 39.0°C - <= 40.0°C | 5 | 2
  Related temperature | 33 | 7

19. Secondary Outcome: Number of Days With Any Grade of Solicited General Symptoms.
Description: as for outcome 17
Time Frame: During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Population: as for outcome 14
Measure: Mean (Full Range); unit: Days
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 446 | 313
Days
  Arthralgia: number analyzed (Participants) | 247 | 169
  Arthralgia | 2.7 [1.0 to 7.0] | 3.0 [1.0 to 7.0]
  Fatigue | 2.6 [1.0 to 7.0] | 2.7 [1.0 to 7.0]
  Gastrointestinal: number analyzed (Participants) | 125 | 115
  Gastrointestinal | 2.3 [1.0 to 7.0] | 2.6 [1.0 to 7.0]
  Headache: number analyzed (Participants) | 331 | 229
  Headache | 2.2 [1.0 to 7.0] | 2.4 [1.0 to 7.0]
  Myalgia: number analyzed (Participants) | 370 | 200
  Myalgia | 2.4 [1.0 to 7.0] | 2.6 [1.0 to 7.0]
  Shivering: number analyzed (Participants) | 177 | 80
  Shivering | 1.6 [1.0 to 7.0] | 2.3 [1.0 to 7.0]
  Temperature: number analyzed (Participants) | 38 | 13
  Temperature | 1.2 [1.0 to 4.0] | 1.5 [1.0 to 4.0]

20. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Unsolicited Adverse Events (AEs).
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Grade 3 = event that prevented normal, everyday activities. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 21 days (Days 0-20) after the first dose (Year 2008/2009)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 3015 | 3002
Participants
  Any AEs | 428 | 427
  Grade 3 AEs | 48 | 52
  Related AEs | 83 | 58

21. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Unsolicited Adverse Events (AEs).
Description: as for outcome 20
Time Frame: Within 21 days (Days 0-20) after the second dose (Year 2009/2010)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 2462 | 2520
Participants
  Any AEs | 320 | 306
  Grade 3 AEs | 36 | 26
  Related AEs | 42 | 20

22. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Unsolicited AEs With Medically Attended Visit
Description: For each solicited and unsolicited symptom the subject experienced, the subjects were asked if they received medical attention defined as hospitalisation, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason. Grade 3 = event that prevented normal everyday activities. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 180 days (Days 0-179) after the first dose (Year 2008/2009)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 3015 | 3002
Participants
  Any AEs | 1018 | 996
  Grade 3 AEs | 223 | 211
  Related AEs | 16 | 7

23. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Unsolicited AEs With Medically Attended Visit.
Description: as for outcome 22
Time Frame: Within 180 days (Days 0-179) after the second dose (Year 2009/2010)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 2462 | 2520
Participants
  Any AEs | 849 | 864
  Grade 3 AEs | 158 | 154
  Related AEs | 7 | 5

24. Secondary Outcome: Serum Hemagglutination-inhibition (HI) Antibody Titer Against Each of the 3 Vaccine Influenza Strains.
Description: Vaccine strains assessed were A/Brisbane/59/2077, A/Uruguay/716/2007 and B/Brisbane/3/2007. Titers were expressed as geometric mean titers calculated on all subjects in the immunogenicity subset of subjects.
Time Frame: At Days 0 (pre-vaccination Dose 1) and 21 (post-vaccination Dose 1) of the first year (2008/2009) of the study
Population: The One-Dose According-To-Protocol cohort for immunogenicity included evaluable subjects for whom data concerning immunogenicity outcome measures were available in terms of antibodies against at least one study vaccine antigen component at Day 21 of the first year of the study.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 2422 | 2408
Titers
  A/Brisbane [Day 0]: number analyzed (Participants) | 2417 | 2397
  A/Brisbane [Day 0] | 15.5 [14.9 to 16.1] | 15.3 [14.7 to 16.0]
  A/Brisbane [Day 21] | 89.1 [85.2 to 93.2] | 69.9 [66.5 to 73.4]
  A/Uruguay [Day 0]: number analyzed (Participants) | 2417 | 2397
  A/Uruguay [Day 0] | 17.4 [16.6 to 18.3] | 17.4 [16.5 to 18.2]
  A/Uruguay [Day 21] | 285.6 [270.6 to 301.4] | 172.3 [162.7 to 182.5]
  B/Brisbane [Day 0]: number analyzed (Participants) | 2416 | 2397
  B/Brisbane [Day 0] | 85.3 [81.2 to 89.7] | 82.4 [78.3 to 86.7]
  B/Brisbane [Day 21] | 633.5 [609.9 to 658.0] | 484.8 [465.1 to 505.4]

25. Secondary Outcome: Serum Hemagglutination-inhibition (HI) Antibody Titer Against Each of the 3 Vaccine Influenza Strains
Description: as for outcome 24
Time Frame: At Days 0 (pre-vaccination Dose 2) and 21 (post-vaccination Dose 2) of the second year (2009/2010) of the study
Population: The Two-Dose According-To-Protocol cohort for immunogenicity included evaluable subjects for whom data concerning immunogenicity outcome measures were available in terms of antibodies against at least one study vaccine antigen component at Day 21 of the second year of the study.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 1938 | 1953
Titers
  A/Brisbane [Day 0]: number analyzed (Participants) | 1932 | 1942
  A/Brisbane [Day 0] | 23.9 [22.9 to 25.0] | 24.3 [23.2 to 25.5]
  A/Brisbane [Day 21]: number analyzed (Participants) | 1936 | 1952
  A/Brisbane [Day 21] | 76.9 [73.6 to 80.4] | 70.5 [67.1 to 74.0]
  A/Uruguay [Day 0]: number analyzed (Participants) | 1932 | 1942
  A/Uruguay [Day 0] | 57.8 [54.5 to 61.3] | 46.5 [43.9 to 49.4]
  A/Uruguay [Day 21]: number analyzed (Participants) | 1937 | 1953
  A/Uruguay [Day 21] | 256.8 [245.3 to 268.9] | 162.0 [153.9 to 170.4]
  B/Brisbane [Day 0]: number analyzed (Participants) | 1933 | 1942
  B/Brisbane [Day 0] | 58.6 [55.6 to 61.8] | 56.6 [53.6 to 59.7]
  B/Brisbane [Day 21] | 199.2 [190.8 to 207.9] | 171.3 [163.6 to 179.4]

26. Secondary Outcome: Serum Hemagglutination-inhibition (HI) Antibody Titer Against Each of the 3 Vaccine Influenza Strains.
Description: Vaccine strains assessed were A/Brisbane/59/2077, A/Uruguay/716/2007 and B/Brisbane/3/2007. Titers were expressed as geometric mean titers calculated on all subjects for 600 subjects in the persistence subset only.
Time Frame: At Days 0 (pre-vaccination Dose 1), 21 (post-vaccination Dose 1) and 180 (post-vaccination Dose 1) of the first year (2008/2009) of the study
Population: The One-Dose According-To-Protocol cohort for persistence included evaluable subjects for whom data concerning immunogenicity outcome measures were available in terms of antibodies against at least one study vaccine antigen component at Day 180 of the first year of the study.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 268 | 267
Titers
  A/Brisbane [Day 0]: number analyzed (Participants) | 268 | 265
  A/Brisbane [Day 0] | 15.4 [13.7 to 17.4] | 13.9 [12.4 to 15.6]
  A/Brisbane [Day 21] | 75.4 [66.3 to 85.9] | 64.5 [55.7 to 74.7]
  A/Brisbane [Day 180] | 30.4 [26.8 to 34.4] | 28.1 [24.8 to 31.8]
  A/Uruguay [Day 0]: number analyzed (Participants) | 268 | 265
  A/Uruguay [Day 0] | 19.3 [16.5 to 22.6] | 17.8 [15.3 to 20.7]
  A/Uruguay [Day 21] | 275.0 [233.1 to 324.5] | 165.0 [139.0 to 195.9]
  A/Uruguay [Day 180] | 97.7 [82.3 to 116.0] | 64.0 [53.7 to 76.3]
  B/Brisbane [Day 0]: number analyzed (Participants) | 268 | 265
  B/Brisbane [Day 0] | 89.3 [76.6 to 104.2] | 83.8 [72.3 to 97.1]
  B/Brisbane [Day 21] | 573.4 [517.5 to 635.3] | 478.5 [422.4 to 541.9]
  B/Brisbane [Day 180] | 274.6 [246.5 to 305.9] | 262.3 [234.7 to 293.1]

27. Secondary Outcome: Serum Hemagglutination-inhibition (HI) Antibody Titer Against Each of the 3 Vaccine Influenza Strains.
Description: as for outcome 26
Time Frame: At Days 0 (pre-vaccination Dose 2), 21 (post-vaccination Dose 2) and 180 (post-vaccination Dose 2) of the second year (2009/2010) of the study
Population: The Two-Dose According-To-Protocol cohort for persistence included evaluable subjects for whom data concerning immunogenicity outcome measures were available in terms of antibodies against at least one study vaccine antigen component at Day 180 of the second year of the study.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FluNG Group | Fluarix Group
Number analyzed (Participants) | 189 | 177
Titers
  A/Brisbane [Day 0]: number analyzed (Participants) | 188 | 177
  A/Brisbane [Day 0] | 23.4 [20.3 to 27.1] | 25.0 [21.3 to 29.3]
  A/Brisbane [Day 21]: number analyzed (Participants) | 188 | 176
  A/Brisbane [Day 21] | 80.0 [69.4 to 92.2] | 75.0 [63.4 to 88.6]
  A/Brisbane [Day 180] | 28.5 [24.7 to 32.8] | 27.3 [23.5 to 31.7]
  A/Uruguay [Day 0]: number analyzed (Participants) | 188 | 177
  A/Uruguay [Day 0] | 68.9 [56.2 to 84.5] | 54.2 [44.1 to 66.5]
  A/Uruguay [Day 21]: number analyzed (Participants) | 188 | 176
  A/Uruguay [Day 21] | 300.6 [254.0 to 355.7] | 195.6 [165.5 to 231.2]
  A/Uruguay [Day 180] | 105.7 [87.9 to 127.2] | 63.6 [53.0 to 76.3]
  B/Brisbane [Day 0] | 58.5 [48.8 to 70.1] | 56.1 [47.0 to 67.0]
  B/Brisbane [Day 21]: number analyzed (Participants) | 189 | 176
  B/Brisbane [Day 21] | 225.1 [195.5 to 259.1] | 191.0 [161.3 to 226.3]
  B/Brisbane [Day 180] | 122.9 [106.5 to 141.7] | 111.6 [95.8 to 130.0]

28. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Each of the 3 Vaccine Influenza Strains
Description: In the lot-to-lot subset of subject in the FluGN Group. Vaccine strains assessed were A/Brisbane/59/2077, A/Uruguay/716/2007 and B/Brisbane/3/2007. Seroconversion is defined as the number of subjects with pre-vaccination HI titer (Day 0) < 1:10 and post-vaccination titer (Day 21) ≥ 1:40 or a pre-vaccination HI titer (Day 0) ≥ 1:10 and fold-increase (post/pre) ≥ 4.
Time Frame: At Day 21 of the first year (2008/2009) of the study.
Population: The One-Dose According-To-Protocol immunogenicity cohort for the lot-to-lot consistency subset included all subjects from the One-Dose ATP cohort for immunogenicity included in the lot-to-lot subset.
Measure: Count of Participants; unit: Participants
Arm/Group | FluNG Lot 1 Group | FluNG Lot 2 Group | FluNG Lot 3 Group
Number analyzed (Participants) | 539 | 536 | 532
Participants
  A/Brisbane | 307 | 298 | 310
  A/Uruguay | 471 | 461 | 455
  B/Brisbane | 389 | 350 | 363

ADVERSE EVENTS:
Time Frame: Solicited symptoms: During the 7-day post-vaccination period the first year (2008/2009) and the second year (2009/2010). SAEs: During the entire study period (during the 365 days of follow-up after each vaccination at Year 2008/2009 and Year 2009/2010)
Arm/Group | FluNG Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 4071/21893 | 4066/21802
Other Adverse Events (participants affected / at risk) | 1999/3015 | 1360/3002
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FluNG Group (N=21893) | Fluarix Group (N=21802)
Pneumonia (Infections and infestations) | 228 | 226
Atrial fibrillation (Cardiac disorders) | 211 | 178
Cerebrovascular accident (Nervous system disorders) | 196 | 180
Myocardial infarction (Cardiac disorders) | 169 | 167
Cardiac failure congestive (Cardiac disorders) | 147 | 153
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 141 | 128
Urinary tract infection (Infections and infestations) | 129 | 111
Cardiac failure (Cardiac disorders) | 98 | 102
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 87 | 108
Coronary artery disease (Cardiac disorders) | 90 | 75
Hypertension (Vascular disorders) | 82 | 83
Angina pectoris (Cardiac disorders) | 77 | 75
Myocardial ischaemia (Cardiac disorders) | 64 | 62
Transient ischaemic attack (Nervous system disorders) | 69 | 57
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 57 | 60
Anaemia (Blood and lymphatic system disorders) | 48 | 64
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 47 | 61
Renal failure acute (Renal and urinary disorders) | 60 | 45
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 61 | 43
Acute myocardial infarction (Cardiac disorders) | 38 | 59
Syncope (Nervous system disorders) | 54 | 43
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 48 | 46
Cholelithiasis (Hepatobiliary disorders) | 44 | 45
Femoral neck fracture (Injury, poisoning and procedural complications) | 35 | 53
Chest pain (General disorders) | 42 | 45
Sepsis (Infections and infestations) | 41 | 45
Cholecystitis (Hepatobiliary disorders) | 40 | 43
Gastroenteritis (Infections and infestations) | 35 | 47
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 44 | 35
Femur fracture (Injury, poisoning and procedural complications) | 34 | 45
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 32 | 37
Diverticulitis (Infections and infestations) | 31 | 34
Inguinal hernia (Gastrointestinal disorders) | 37 | 26
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 | 38
Arrhythmia (Cardiac disorders) | 35 | 26
Cardiac arrest (Cardiac disorders) | 33 | 28
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 27 | 31
Hip fracture (Injury, poisoning and procedural complications) | 23 | 34
Renal failure chronic (Renal and urinary disorders) | 27 | 30
Cellulitis (Infections and infestations) | 29 | 27
Bronchopneumonia (Infections and infestations) | 26 | 29
Death (General disorders) | 28 | 27
Humerus fracture (Injury, poisoning and procedural complications) | 19 | 35
Renal failure (Renal and urinary disorders) | 26 | 27
Arteriosclerosis (Vascular disorders) | 22 | 30
Sudden death (General disorders) | 34 | 18
Asthma (Respiratory, thoracic and mediastinal disorders) | 33 | 17
Dehydration (Metabolism and nutrition disorders) | 24 | 25
Erysipelas (Infections and infestations) | 28 | 21
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 19 | 29
Hypertensive crisis (Vascular disorders) | 26 | 21
Cerebrovascular disorder (Nervous system disorders) | 24 | 21
Ischaemic stroke (Nervous system disorders) | 17 | 28
Depression (Psychiatric disorders) | 24 | 20
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 18 | 26
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 19 | 24
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 22 | 20
Gastritis (Gastrointestinal disorders) | 20 | 22
Circulatory collapse (Vascular disorders) | 23 | 18
Hypoglycaemia (Metabolism and nutrition disorders) | 23 | 18
Cholecystitis acute (Hepatobiliary disorders) | 23 | 17
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 19
Bradycardia (Cardiac disorders) | 18 | 20
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 22 | 15
Deep vein thrombosis (Vascular disorders) | 13 | 24
Cataract (Eye disorders) | 16 | 20
Diabetes mellitus (Metabolism and nutrition disorders) | 18 | 18
Pancreatitis acute (Gastrointestinal disorders) | 18 | 18
Angina unstable (Cardiac disorders) | 17 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 20
Lobar pneumonia (Infections and infestations) | 16 | 19
Rib fracture (Injury, poisoning and procedural complications) | 21 | 14
Toxicity to various agents (Injury, poisoning and procedural complications) | 17 | 18
Cerebral infarction (Nervous system disorders) | 23 | 11
Gastric ulcer (Gastrointestinal disorders) | 16 | 18
Intestinal obstruction (Gastrointestinal disorders) | 15 | 19
Nephrolithiasis (Renal and urinary disorders) | 14 | 20
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 15 | 19
Pyelonephritis (Infections and infestations) | 21 | 13
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 21
Radius fracture (Injury, poisoning and procedural complications) | 13 | 20
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 19 | 14
Vertigo (Ear and labyrinth disorders) | 14 | 19
Appendicitis (Infections and infestations) | 15 | 17
Contusion (Injury, poisoning and procedural complications) | 20 | 12
Peripheral arterial occlusive disease (Vascular disorders) | 19 | 13
Atrial flutter (Cardiac disorders) | 14 | 16
Upper respiratory tract infection (Infections and infestations) | 13 | 17
Ankle fracture (Injury, poisoning and procedural complications) | 14 | 15
Pancreatitis (Gastrointestinal disorders) | 18 | 11
Aortic aneurysm (Vascular disorders) | 13 | 15
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 13
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 16 | 12
Urinary retention (Renal and urinary disorders) | 13 | 15
Atrioventricular block (Cardiac disorders) | 11 | 16
Hypotension (Vascular disorders) | 14 | 13
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 12
Concussion (Injury, poisoning and procedural complications) | 10 | 16
Upper limb fracture (Injury, poisoning and procedural complications) | 9 | 17
Epilepsy (Nervous system disorders) | 14 | 11
Ileus (Gastrointestinal disorders) | 14 | 11
Small intestinal obstruction (Gastrointestinal disorders) | 13 | 12
Spinal compression fracture (Injury, poisoning and procedural complications) | 14 | 11
Wrist fracture (Injury, poisoning and procedural complications) | 15 | 10
Acute coronary syndrome (Cardiac disorders) | 6 | 18
Bile duct stone (Hepatobiliary disorders) | 15 | 9
Constipation (Gastrointestinal disorders) | 11 | 13
Mitral valve incompetence (Cardiac disorders) | 14 | 10
Multi-organ failure (General disorders) | 9 | 15
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Septic shock (Infections and infestations) | 6 | 18
Carotid artery stenosis (Nervous system disorders) | 13 | 10
Duodenal ulcer (Gastrointestinal disorders) | 15 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Haematoma (Vascular disorders) | 15 | 8
Peritonitis (Gastrointestinal disorders) | 12 | 11
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 13
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 9
Colitis (Gastrointestinal disorders) | 8 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 9
Peripheral vascular disorder (Vascular disorders) | 11 | 11
Aortic valve stenosis (Cardiac disorders) | 13 | 8
Gangrene (Infections and infestations) | 10 | 11
Iron deficiency anaemia (Blood and lymphatic system disorders) | 7 | 14
Sick sinus syndrome (Cardiac disorders) | 10 | 11
Abdominal pain (Gastrointestinal disorders) | 13 | 7
Atrioventricular block complete (Cardiac disorders) | 9 | 11
Colonic polyp (Gastrointestinal disorders) | 11 | 9
Hepatic cirrhosis (Hepatobiliary disorders) | 11 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 9 | 11
Pelvic fracture (Injury, poisoning and procedural complications) | 9 | 11
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 8 | 12
Subdural haematoma (Injury, poisoning and procedural complications) | 5 | 15
Supraventricular tachycardia (Cardiac disorders) | 7 | 13
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 | 9
Cardiac death (General disorders) | 11 | 8
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 9 | 10
Sudden cardiac death (General disorders) | 12 | 7
Vascular dementia (Nervous system disorders) | 12 | 7
Aortic stenosis (Vascular disorders) | 11 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 12
Cerebral ischaemia (Nervous system disorders) | 9 | 9
Road traffic accident (Injury, poisoning and procedural complications) | 9 | 9
Cystitis (Infections and infestations) | 5 | 12
Diarrhoea (Gastrointestinal disorders) | 8 | 9
Facial bones fracture (Injury, poisoning and procedural complications) | 9 | 8
Gastritis erosive (Gastrointestinal disorders) | 9 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 10
Head injury (Injury, poisoning and procedural complications) | 9 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 9
Left ventricular failure (Cardiac disorders) | 9 | 8
Non-cardiac chest pain (General disorders) | 9 | 8
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 12 | 5
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9
Tachyarrhythmia (Cardiac disorders) | 9 | 8
Venous thrombosis (Vascular disorders) | 9 | 8
Coronary artery stenosis (Cardiac disorders) | 7 | 9
Diverticulum (Gastrointestinal disorders) | 7 | 9
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 7 | 9
Haematuria (Renal and urinary disorders) | 8 | 8
Herpes zoster (Infections and infestations) | 7 | 9
Hiatus hernia (Gastrointestinal disorders) | 5 | 11
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 6 | 10
Joint dislocation (Injury, poisoning and procedural complications) | 5 | 11
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 7 | 9
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 7
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 6
Respiratory tract infection (Infections and infestations) | 7 | 9
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 8 | 8
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 8 | 8
Arrhythmia supraventricular (Cardiac disorders) | 11 | 4
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 7
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 8
Spinal fracture (Injury, poisoning and procedural complications) | 6 | 9
Ventricular fibrillation (Cardiac disorders) | 8 | 7
Wound infection (Infections and infestations) | 8 | 7
Calculus ureteric (Renal and urinary disorders) | 10 | 4
Colitis ischaemic (Gastrointestinal disorders) | 3 | 11
Laceration (Injury, poisoning and procedural complications) | 8 | 6
Lower limb fracture (Injury, poisoning and procedural complications) | 8 | 6
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 7
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 5
Cardiopulmonary failure (Cardiac disorders) | 7 | 6
Cerebral haemorrhage (Nervous system disorders) | 9 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 6 | 7
Dementia (Nervous system disorders) | 4 | 9
Dementia alzheimer's type (Nervous system disorders) | 9 | 4
Dizziness (Nervous system disorders) | 5 | 8
Fall (Injury, poisoning and procedural complications) | 4 | 9
Large intestine perforation (Gastrointestinal disorders) | 8 | 5
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 4
Parkinson's disease (Nervous system disorders) | 8 | 5
Presyncope (Nervous system disorders) | 9 | 4
Staphylococcal infection (Infections and infestations) | 8 | 5
Tendon rupture (Injury, poisoning and procedural complications) | 10 | 3
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 5
Urethral stenosis (Renal and urinary disorders) | 3 | 10
Vestibular disorder (Ear and labyrinth disorders) | 5 | 8
Arteriosclerosis coronary artery (Cardiac disorders) | 6 | 6
Cardiac failure chronic (Cardiac disorders) | 7 | 5
Cardio-respiratory arrest (Cardiac disorders) | 5 | 7
Cardiovascular insufficiency (Cardiac disorders) | 6 | 6
Completed suicide (Psychiatric disorders) | 5 | 7
Coronary artery occlusion (Cardiac disorders) | 6 | 6
Diabetic foot (Metabolism and nutrition disorders) | 5 | 7
Dyspepsia (Gastrointestinal disorders) | 4 | 8
Grand mal convulsion (Nervous system disorders) | 4 | 8
Haemorrhoids (Gastrointestinal disorders) | 7 | 5
Hypersensitivity (Immune system disorders) | 7 | 5
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 7
Reflux oesophagitis (Gastrointestinal disorders) | 3 | 9
Sciatica (Nervous system disorders) | 7 | 5
Thrombophlebitis (Vascular disorders) | 7 | 5
Thrombosis (Vascular disorders) | 4 | 8
Urosepsis (Infections and infestations) | 8 | 4
Calculus bladder (Renal and urinary disorders) | 6 | 5
Cardiac failure acute (Cardiac disorders) | 6 | 5
Cerebral arteriosclerosis (Nervous system disorders) | 7 | 4
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Fibula fracture (Injury, poisoning and procedural complications) | 7 | 4
Glaucoma (Eye disorders) | 3 | 8
Hydronephrosis (Renal and urinary disorders) | 8 | 3
Hypothyroidism (Endocrine disorders) | 4 | 7
Orthostatic hypotension (Vascular disorders) | 5 | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 | 6
Subarachnoid haemorrhage (Nervous system disorders) | 7 | 4
Tibia fracture (Injury, poisoning and procedural complications) | 3 | 8
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Arterial occlusive disease (Vascular disorders) | 4 | 6
Atrioventricular block second degree (Cardiac disorders) | 8 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Brain oedema (Nervous system disorders) | 3 | 7
Cholangitis (Hepatobiliary disorders) | 5 | 5
Delirium (Psychiatric disorders) | 6 | 4
Dysphagia (Gastrointestinal disorders) | 3 | 7
Faecaloma (Gastrointestinal disorders) | 4 | 6
Hyperthyroidism (Endocrine disorders) | 1 | 9
Intermittent claudication (Vascular disorders) | 4 | 6
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 8
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Sinusitis (Infections and infestations) | 3 | 7
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
Traumatic brain injury (Injury, poisoning and procedural complications) | 5 | 5
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
Uterine prolapse (Reproductive system and breast disorders) | 7 | 3
Ventricular tachycardia (Cardiac disorders) | 4 | 6
Vertigo positional (Ear and labyrinth disorders) | 2 | 8
Abdominal hernia (Gastrointestinal disorders) | 6 | 3
Angioedema (Skin and subcutaneous tissue disorders) | 4 | 5
Aortic valve incompetence (Cardiac disorders) | 3 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 4
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 5 | 4
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Haemorrhagic stroke (Nervous system disorders) | 5 | 4
Hand fracture (Injury, poisoning and procedural complications) | 4 | 5
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 8
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Oesophagitis (Gastrointestinal disorders) | 5 | 4
Osteomyelitis (Infections and infestations) | 2 | 7
Ovarian cyst (Reproductive system and breast disorders) | 4 | 5
Pancreatitis chronic (Gastrointestinal disorders) | 6 | 3
Peripheral ischaemia (Vascular disorders) | 5 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Umbilical hernia (Gastrointestinal disorders) | 4 | 5
Urinary bladder polyp (Renal and urinary disorders) | 3 | 6
Vertebrobasilar insufficiency (Nervous system disorders) | 4 | 5
Arterial thrombosis limb (Vascular disorders) | 4 | 4
Asthenia (General disorders) | 5 | 3
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Calculus urinary (Renal and urinary disorders) | 2 | 6
Cardiogenic shock (Cardiac disorders) | 6 | 2
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Clostridial infection (Infections and infestations) | 2 | 6
Clostridium difficile colitis (Infections and infestations) | 5 | 3
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Confusional state (Psychiatric disorders) | 4 | 4
Convulsion (Nervous system disorders) | 3 | 5
Cystitis haemorrhagic (Renal and urinary disorders) | 5 | 3
Diverticular perforation (Gastrointestinal disorders) | 2 | 6
Diverticulum intestinal (Gastrointestinal disorders) | 6 | 2
Encephalopathy (Nervous system disorders) | 6 | 2
Foot fracture (Injury, poisoning and procedural complications) | 5 | 3
Forearm fracture (Injury, poisoning and procedural complications) | 7 | 1
Goitre (Endocrine disorders) | 5 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 5
Infection (Infections and infestations) | 2 | 6
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Peptic ulcer (Gastrointestinal disorders) | 5 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pyrexia (General disorders) | 3 | 5
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Retinal detachment (Eye disorders) | 2 | 6
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Tachycardia (Cardiac disorders) | 3 | 5
Ventricular extrasystoles (Cardiac disorders) | 4 | 4
Vomiting (Gastrointestinal disorders) | 5 | 3
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Anaphylactic reaction (Immune system disorders) | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Brain contusion (Injury, poisoning and procedural complications) | 2 | 5
Candidiasis (Infections and infestations) | 5 | 2
Cholecystitis infective (Infections and infestations) | 4 | 3
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Coronary artery insufficiency (Cardiac disorders) | 2 | 5
Device dislocation (General disorders) | 2 | 5
Duodenitis (Gastrointestinal disorders) | 3 | 4
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Gastric haemorrhage (Gastrointestinal disorders) | 5 | 2
Gastroenteritis norovirus (Infections and infestations) | 3 | 4
Gastroenteritis viral (Infections and infestations) | 3 | 4
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4 | 3
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2
Hypertensive heart disease (Cardiac disorders) | 3 | 4
Hypovolaemic shock (Vascular disorders) | 5 | 2
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Multiple injuries (Injury, poisoning and procedural complications) | 3 | 4
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Nausea (Gastrointestinal disorders) | 5 | 2
Oedema peripheral (General disorders) | 4 | 3
Oesophageal stenosis (Gastrointestinal disorders) | 3 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 | 3
Overdose (Injury, poisoning and procedural complications) | 3 | 4
Parkinsonism (Nervous system disorders) | 6 | 1
Pericarditis (Cardiac disorders) | 2 | 5
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Prostatitis (Reproductive system and breast disorders) | 3 | 4
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 6
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 | 4
Ulna fracture (Injury, poisoning and procedural complications) | 3 | 4
Uterine polyp (Reproductive system and breast disorders) | 4 | 3
Varicose vein (Vascular disorders) | 6 | 1
Biliary colic (Hepatobiliary disorders) | 3 | 3
Bladder neck obstruction (Renal and urinary disorders) | 1 | 5
Brain stem infarction (Nervous system disorders) | 3 | 3
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Cachexia (Metabolism and nutrition disorders) | 3 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 | 3
Embolic stroke (Nervous system disorders) | 3 | 3
Escherichia urinary tract infection (Infections and infestations) | 6 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 4
Gastroduodenal ulcer (Gastrointestinal disorders) | 4 | 2
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 3 | 3
Gout (Metabolism and nutrition disorders) | 6 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 5
Ileus paralytic (Gastrointestinal disorders) | 5 | 1
Infected skin ulcer (Infections and infestations) | 2 | 4
Infective exacerbation of chronic obstructive airways diseas (Infections and infestations) | 3 | 3
Injury (Injury, poisoning and procedural complications) | 3 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 4 | 2
Intestinal polyp (Gastrointestinal disorders) | 5 | 1
Localised infection (Infections and infestations) | 3 | 3
Lower respiratory tract infection (Infections and infestations) | 2 | 4
Lung infection (Infections and infestations) | 1 | 5
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 | 4
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Pain (General disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Pharyngitis (Infections and infestations) | 2 | 4
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 5
Postoperative wound infection (Infections and infestations) | 2 | 4
Pyelonephritis acute (Infections and infestations) | 4 | 2
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2
Vascular encephalopathy (Nervous system disorders) | 2 | 4
Venous thrombosis limb (Vascular disorders) | 3 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FluNG Group (N=3015) | Fluarix Group (N=3002)
Pain (General disorders) | 1225 | 477 — During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Redness (General disorders) | 240 | 66 — During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Swelling (General disorders) | 189 | 40 — During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Pain (General disorders) | 998 | 440 — During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Redness (General disorders) | 212 | 54 — During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Swelling (General disorders) | 173 | 38 — During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Arthralgia (General disorders) | 391 | 239 — During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Fatigue (General disorders) | 646 | 417 — During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Gastrointestinal (General disorders) | 197 | 165 — During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Headache (General disorders) | 474 | 333 — During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Myalgia (General disorders) | 547 | 302 — During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Shivering (General disorders) | 245 | 80 — During the 7-day (Days 0-6) post-vaccination period, the first year (2008/2009)
Arthralgia (General disorders) | 258 | 176 — During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Fatigue (General disorders) | 457 | 318 — During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Gastrointestinal (General disorders) | 137 | 124 — During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Headache (General disorders) | 342 | 237 — During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Myalgia (General disorders) | 380 | 209 — During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)
Shivering (General disorders) | 189 | 88 — During the 7-day (Days 0-6) post-vaccination period, the second year (2009/2010)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.